CLINICAL TRIAL: NCT05597124
Title: Determinants of Individual Differences in the Efficacy of Aerobic Exercise to Improve Brain Health and Reduce Alzheimer's Disease Risk in Older African Americans
Brief Title: Exercise to Improve Brain Health in Older African Americans
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Göteborg University (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Mark A. Gluck, PhD, Principal Investigator, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro2022001256
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Aging; Alzheimer Disease; Healthy Aging; Cognitive Change
MeSH Terms: conditions — Alzheimer Disease | interventions — Pliability

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardio-Dance Fitness (Experimental): This is the experimental group. Participants will meet three times a week for dance classes for approximately 60 minutes per session, over 24 weeks (approximately 6 months).
  Interventions: Behavioral: Cardio-Dance Fitness
- Strength, Flexibility & Balance (Active Comparator): This is the active control group. Participants will meet three times a week for strength, flexibility, and balance exercises for approximately 60 minutes per session, over 24 weeks (approximately 6 months).
  Interventions: Behavioral: Strength, Flexibility & Balance

INTERVENTIONS:
Behavioral: Cardio-Dance Fitness — This is an aerobic cardio-dance fitness exercise class in a social context with aerobic intensity assessed by heart rate monitoring throughout the class. Participants will meet three times a week for approximately 60 minutes per session, over 24 weeks (approximately 6 months).
  Other Names: CDF
  Arms: Cardio-Dance Fitness
Behavioral: Strength, Flexibility & Balance — This intervention will serve as a stringent, structurally equivalent, active comparator to the CDF intervention, identical in duration, frequency, and social contact except for the content of this non-aerobic intervention. SFB will involve non-aerobic activity with strength, flexibility, and balance training.
  Other Names: SFB
  Arms: Strength, Flexibility & Balance

SUMMARY:
The goal of this clinical trial is to test the effects of different types of exercise on brain health and Alzheimer's risk in older African Americans.

Specifically, the main question[s] it aims to answer are:

* What is the effect of a Cardio-Dance Fitness (CDF) vs. a Strength, Flexibility, and Balance (SFB) intervention on a cognitive marker of Alzheimer's risk, generalization?
* What is the effect of the CDF vs. SFB intervention on a fMRI biomarker of Alzheimer's, neural flexibility, and do improvements in neural flexibility mediate improvements in generalization?
* Do ABCA7 genotypic variations moderate the efficacy of the CDF vs. SFB intervention for reducing Alzheimer's risk?

Participants will undergo-- at baseline and post-test-- health assessments, cognitive tests, and structural and functional magnetic resonance imaging (fMRI), and a blood-draw to assess Alzheimer's risk biomarker levels.

DETAILED DESCRIPTION:
Older African Americans-especially those with lower income and those living in urban neighborhoods- have a greater risk of Alzheimer's disease (AD) compared to the general population. This health disparity is attributable, in part, to modifiable factors including insufficient levels of aerobic exercise. However, not everyone gains the same degree of neuroprotection from exercise. For the proposed project, the investigators plan to investigate genetic risk as a novel source of response heterogeneity to exercise interventions in African Americans. Previously, the investigators demonstrated that five months of twice-weekly cardio-dance exercise can increase the dynamic rearrangement (or "neural flexibility") of resting-state networks within the medial temporal lobe (MTL), one of the earliest brain regions impacted by AD. Moreover, this improved neural flexibility mediates intervention-related improvements in generalization, the ability to apply past learning to novel task demands. Given our earlier findings that generalization is impaired in preclinical AD, these results suggest a novel circuit-level mechanism, MTL neural flexibility, through which exercise may reduce risk for dementia. Moreover, the investigators discovered that the cognitive benefits of exercise in older African Americans are diminished in those with a risk variant of the ABCA7 (rs3764650) gene. Two key limitations to our previous exercise studies were: (1) interventions limited to two 60-minute classes/week, below the recommended 150 minutes/week, and (2) too few participants to evaluate the effect of ABCA7 on exercise-induced changes on neural flexibility. The investigators propose to recruit 280 sedentary older African Americans, ages 60 and above, to be randomized to one of two equally engaging six-month interventions, a Cardio Dance Fitness (CDF) intervention, and a Strength, Flexibility, & Balance active control. All participants will undergo-at enrollment and post-intervention-health assessments, cognitive tests, and structural and functional magnetic resonance imaging (fMRI), and a blood-draw to assess amyloid (Aβ 42/40) and tau (p-tau231, p-tau181). This will enable us to test: 1) the effect of the CDF intervention on a cognitive marker of AD risk, generalization; 2) the effect of the CDF intervention on a fMRI biomarker of AD, neural flexibility, and determine whether improvements in neural flexibility mediate improvements in generalization; and 3) whether ABCA7 genotypic variations moderate the efficacy of the CDF intervention for reducing AD risk. Impact: This work lays the foundation for future larger clinical trials to develop personalized exercise prescriptions for older African Americans with varying genetic, health, and social-determinant risk profiles, so as to optimize the impact of this low-cost non-pharmaceutical intervention for improving their brain health.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as either African American or Black;
* be age 60 or older;
* able to speak, read, and understand English;
* available over the study period; independently ambulatory (i.e., not needing a wheelchair, walker, or cane);
* meet criteria for low levels of physical activity (less than 60 minutes per week) based on the International Physical Activity Questionnaire (IPAQ-short version);
* scoring 28-35 (inclusive) on the Telephone Interview for Cognitive Status Modified (sensitivity [43%], specificity [94%] for lower threshold; sensitivity [93%], specificity [42%] for upper threshold)55.
* scoring 20-26 (inclusive) on the Montreal Cognitive Assessment (MoCA) during the in-person screening
* have clearance to participate from their primary care physician, with oversight of all our patient health under the guidance of our physician-scientist Co-I, William Hu, Chief of Cognitive Neurology at Rutgers.

Exclusion Criteria:

* color-blindness (because some of our tasks utilize color as a cue);
* any diagnosed neurological disorder (including headaches and peripheral neuropathy); diagnosed or self-reported non-neurological conditions that likely affect MTL outcomes, such as, major depressive disorder (or a Geriatric Depression Scale-Short Form score ≥ 5), schizophrenia, delusional disorder, schizoaffective disorder or significant psychiatric symptoms that could impair the completion of the study (e.g., psychosis), substance-related and addictive disorders (or treatment in past five years), chemotherapy or radiation treatment for cancers, planning to undergo general anesthesia during the study period;
* exercise contraindications, such as, orthopedic complications, myocardial infarction, coronary artery bypass grafting, angioplasty or other cardiac condition in the past year, current treatment for congestive heart failure, angina, uncontrolled arrhythmia, deep vein thrombosis (DVT) or another cardiovascular event, and uncontrolled hypertension with resting systolic or diastolic blood pressures > 180/110 mmHg.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Generalization Performance on the Concurrent Discrimination and Transfer Task | Changes from baseline to six months
  The Concurrent Discrimination and Transfer Task (a task that indexes generalization, the ability to apply past learning to novel task demands) will be administered at baseline, and then following the intervention (6-months). The main outcome from this task is the number transfer errors. A higher score indicates worse generalization.
Generalization Performance on the Acquired Equivalence Task | Changes from baseline to six months
  The Acquired Equivalence Task (a task that indexes generalization, the ability to apply past learning to novel task demands) will be administered at baseline, and then following the intervention (6-months). The main outcome from this task is generalization accuracy. A higher score indicates better generalization.
Medial Temporal Lobe Neural Flexibility | Changes from baseline to six months
  Medial Temporal Lobe Neural Flexibility is a measure of synchrony via fMRI resting-state analyses in the hippocampus and other medial temporal lobe brain regions for encoding new memories. Flexibility is quantified as the number of times a node displayed a change in community assignment, normalized by the total possible number of changes; this will be computed for each of our seven regions of interest in the medial temporal lobe. A higher score indicates greater flexibility.
  The flexibility of the MTL network as a whole was then computed as the mean flexibility over all nodes.

OTHER OUTCOMES:
Exploratory Outcome: AB 42/40 | Changes from baseline to six months
  The ratio of 42 to 40 amino acid-long amyloid β, a marker of plaque pathology, will be examined as an exploratory outcome. Lower values indicate more AB 42/40 pathology.
Exploratory Outcome: p-tau181 | Changes from baseline to six months
  Phosphorylated tau 181, a marker of AD-related tau phosphorylation and secretion, will be examined as an exploratory outcome. Higher values indicate more tau pathology.
Exploratory Outcome: p-tau231 | Changes from baseline to six months
  Phosphorylated tau 231, a marker of AD-related tau phosphorylation and secretion, will be examined as an exploratory outcome. Higher values indicate more tau pathology.
Exploratory Outcome: Neurofilament-light Chain | Changes from baseline to six months
  Neurofilament-light chain (NfL) is a neuronal cytoplasmic protein; its levels increase in plasma and cerebrospinal fluid proportional to the degree of axonal damage in a variety of neurological disorders, including Alzheimer's disease. Higher values indicate greater axonal damage.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Gluck, PhD, Principal Investigator — Rutgers, The State University of New Jersey - Newark campus
Locations (1):
- Rutgers, The State University of New Jersey - Newark campus, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make the data and associated documentation available to users only under a Data-Sharing Agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: All data will be made available to share with the public after de-identification and following a grace period of six months post-grant completion to allow the PI and team to publish results from the research first.
Access Criteria: Data requests will be approved by the Principal Investigator and Co-Investigators. Requests can be made by completing a data request form.

REFERENCES:
- [Background] Gluck MA, Gills JL, Fausto BA, Malin SK, Duberstein PR, Erickson KI, Hu L. Examining the efficacy of a cardio-dance intervention on brain health and the moderating role of ABCA7 in older African Americans: a protocol for a randomized controlled trial. Front Aging Neurosci. 2023 Nov 21;15:1266423. doi: 10.3389/fnagi.2023.1266423. eCollection 2023. PMID 38076534

DOCUMENTS (1):
  • Informed Consent Form (2024-07-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT05597124/ICF_001.pdf